CLINICAL TRIAL: NCT00974896
Title: A Phase 1b Study of AMG 479 With Biologics or Chemotherapy in Adult Subjects With Advanced Solid Tumors
Brief Title: QUILT-2.016: Study of AMG 479 With Biologics or Chemotherapy for Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060134; QUILT-2.016 (Other: NantCell, Inc.)
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Advanced Malignancy; Advanced Solid Tumors; Cancer; Solid Tumors; Tumors
Keywords: Advanced Solid Tumors; AMG 479; Amgen; Oncology; Phase 1b
MeSH Terms: conditions — Neoplasms | interventions — ganitumab

ARMS (2):
- AMG 479 + Sorafenib cohorts (Experimental): The aim is to determine the safety, tolerability and PK of AMG 479 with sorafenib. AMG 479 will be given bi-weekly; sorafenib will be given daily.
  Interventions: Drug: AMG 479
- AMG 479 + Erlotinib cohorts (Experimental): The aim is to determine the safety, tolerability and PK of AMG 479 with erlotinib. AMG 479 will be given bi-weekly; erlotinib will be given daily.
  Interventions: Drug: AMG 479

INTERVENTIONS:
Drug: AMG 479 — AMG 479 is a fully human IgG1 monoclonal antibody that inhibits IGF-1R signalling. AMG 479 (6mg/kg or 12mg/kg) will be given IV every 2 weeks in combination with sorafenib (400 mg po BID) or erlotinib (150 mg po QD).

SUMMARY:
To assess the safety, tolerability, and pharmacokinetic profiles of AMG 479 when used in combination with bevacizumab, sorafenib, panitumumab, erlotinib, or gemcitabine in subjects with advanced solid tumors. Up to 126 subjects may be enrolled. Sorafenib and erlotinib combo cohorts are enrolling. All other combo cohorts are closed to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Competent to comprehend, sign, and date an Institutional Review Board (IRB) approved informed consent form
* Men and women ≥ 18 years old with a pathologically or cytologically documented, advanced solid tumor that is refractory to at least one line of therapy or for whom no standard therapy is available and for which no curative therapy is available, or the subject refuses standard non-curative therapy
* Measurable disease or evaluable disease per World Health Organization (WHO) guidelines
* Eastern Cooperative Oncology Group performance status ≤ 2
* Life expectancy of 3 months as documented by the investigator
* Adequate hematologic, renal and hepatic function

Exclusion Criteria:

* Any co-morbid medical condition that would increase the risk of toxicity in the opinion of Investigator or Sponsor
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Events (CTCAE) grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* Subjects with primary or metastatic central nervous system (CNS) tumors are not allowed to enroll in the sorafenib cohorts. These subjects are allowed to enroll in the remaining cohorts, only if their CNS tumors have been controlled by prior surgery or radiation, and they have been neurologically stable
* History of lymphoma, leukemia, or high-dose chemotherapy with hematopoietic stem cell rescue
* Uncontrolled hypertension [diastolic >100 mmHg or systolic >150 mmHg]; Subjects enrolling in the sorafenib groups must not have diastolic > 85 mmHg nor systolic > 145 mmHg
* Clinically significant ECG changes which obscure the ability to assess the PR, QT, QRS intervals
* Presence of ascites or pleural effusion requiring chronic medical intervention
* Diagnosis of arterial or venous thrombosis within 6 months before enrollment; history of bleeding diathesis
* History of clinically significant hypoglycemia or hyperglycemia in the opinion of the investigator
* Myocardial infarction within 6 months before enrollment, symptomatic congestive heart failure (New York Heart Association >class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* Active peptic ulcer disease
* History of chronic hepatitis
* Subject known to have tested positive for HIV
* Known sensitivity to mammalian derived products
* Hematological function, as follows:
* Absolute neutrophil count (ANC) ≤ 1.5 x 109/L for B, P, S and E cohorts
* Absolute neutrophil count (ANC) ≤ 3 x 109/L for G cohorts
* Platelet count ≤ 100 x 109/L
* Hemoglobin ≤ 9 g/dL
* Renal function, as follows:
* Calculated creatinine clearance < 50 ml/min using the modified Cockroft-Gault equation
* Urinary protein quantitative value of > 30 mg or >1+ on dipstick, unless quantitative protein is < 500 mg in a 24 hour urine sample
* Hepatic function, as follows:
* Aspartate aminotransferase (AST) > 2.5 x upper limit of normal (ULN) (if liver metastases are present, ≥ 5 x ULN)
* Alanine aminotransferase (ALT) > 2.5 x ULN (if liver metastases are present, ≥ 5 x ULN)
* Alkaline phosphatase > 2.0 x ULN (if bone or liver metastases are present, ≥ 5 x ULN)
* Bilirubin > 2.0 x ULN
* Prothrombin time (PT) or partial thromboplastin time (PTT) > 1.5 x ULN
* Treatment with anti-cancer therapy (6 weeks for nitrosoureas and mitomycin C chemotherapies), antibody therapy, retinoid therapy, or hormonal therapy within 4 weeks before study day 1. Prior and concurrent use of hormone replacement therapy or the use of gonadotropin-releasing hormone (GnRH) modulators for prostate cancer are permitted
* Therapeutic or palliative radiation therapy within 4 weeks before enrollment (subjects must have resolution of any significant adverse effects from radiation therapy received prior to 2 weeks before enrollment)
* Concurrent or prior (within 1 week of study Day 1) anticoagulation therapy, except low-dose warfarin (≤ 2 mg/day) for prophylaxis against central venous catheter thrombosis
* Prior participation in clinical drug trials within 4 weeks before enrollment
* For subjects receiving erlotinib, the use of ketoconazole, clarithromycin, voriconazole, troleandomycin, telithromycin, rifabutin, rifapentine, phenytoin, carbamazepine, phenobarbital and St. John's Wort is prohibited
* For subjects receiving sorafenib, use of St. John's Wort, rifampin, phenytoin, carbamazepine, dexamethasone, and phenobarbital (CYP3A inducers) is prohibited
* Type 1 or 2 diabetics are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-12; Primary Completion 2010-09 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety, tolerability, and pharmacokinetic profiles of AMG 479 when used in combination with bevacizumab, sorafenib, panitumumab, erlotinib or gemcitabine in subjects with advanced solid tumors | 3 years

SECONDARY OUTCOMES:
To evaluate pharmacokinetic (PK) profiles of biologics or chemotherapy when used in combination with AMG 479 | 3 years
To evaluate tumor response as assessed by World Health Organization (WHO) criteria | 3 years
To evaluate tumor response as measured by volumetric computed tomography (CT) | 3 years
To evaluate anti-AMG 479 antibody response following AMG 479 administration | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com